CLINICAL TRIAL: NCT06165315
Title: Evaluation of a Group-based Parenting Intervention for Early Childhood Development
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: ChildFund Kenya (Unknown); Conrad N. Hilton Foundation (Other); B&M Consult (Unknown)
Responsible Party: Principal Investigator, Joshua Jeong, Research Associate, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ISERC/JOOTRH/736/23
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Child Development

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parenting Program (Experimental): This community-based group parenting program aims improve caregiver knowledge, attitudes, and practices on nurturing care to ultimate improve early childhood development. A secondary aim of the program is to support caregiver psychosocial wellbeing. The curriculum covers various topics relating to responsive caregiving, early learning, child protection, maternal and child health and nutrition, and caregiver mental health. Intervention will be delivered through existing community group networks. Each parenting group will comprise of 10 caregivers that will be facilitated by trained volunteers.
  Interventions: Behavioral: Parenting program
- Waitlist-Control (No Intervention): Villages in the control group will not immediately receive the parenting program. Instead, they will receive whatever standard of care services are delivered at the community-level (e.g., routine services from community health volunteers that are primarily focused on maternal and child health and nutrition). After endline data collection is completed for the trial, then villages in the control group will receive the parenting program.

INTERVENTIONS:
Behavioral: Parenting program — Villages in the intervention group will receive the parenting program. The parenting program consists of 20 total sessions, whereby groups will meet twice a month for 10 months.
  Arms: Parenting Program

SUMMARY:
This implementation research study aims to evaluate the impact and implementation of a group-based parenting program for improving early child development and caregiver outcomes. This study is enrolling primary caregivers with children 0 to 24 months of age to promote caregiver knowledge and skills about nurturing care for young children and support caregiver psychosocial wellbeing. Parenting groups will leverage existing community group networks and be facilitated by trained volunteers for 20 total sessions (groups will meet twice a month for 10 months). ChildFund Kenya and its community partners will implement the program in Busia and Homabay counties. The research study design will involve a cluster-randomized controlled trial and a qualitative implementation evaluation. This research is being led by Emory University with funding from the Conrad N. Hilton Foundation.

DETAILED DESCRIPTION:
This research has two study components and aims. First, a cluster-randomized controlled trial will be used to quantitatively estimate the effectiveness of the parenting program on early child development and caregiver outcomes. For the research study sample, villages in Busia and Homabay counties were randomly selected and randomly assigned in each county to either the intervention or waitlist control group. Villages in the intervention group will receive the parenting program first, while villages in the control group will receive the program after the completion of the research study. In total, 64 villages have been selected into this study. Then in each village, 10 primary caregivers with children 0-24 months of age will be enrolled into the study for a total of 640 caregiver-child dyads. A caregiver survey and observational assessment of early child development skills will be administered to study participants at baseline and endline to evaluate changes in outcomes between groups over time. Second, and following the completion of the program, qualitative in-depth interviews will be conducted with participants and various stakeholders (e.g., program participants, parenting group facilitators, community health volunteers, ChildFund program staff) to understand their roles and experiences with the parenting program as well as the challenges and successes to inform future implementation. This qualitative implementation evaluation will seek to identify the barriers and facilitators to program impact, quality delivery, scale-up, and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* primary caregiver of a child aged 0-24 months at the time of enrollment
* the household resides within the geographic boundary of the village that was sampled into the research study
* primary caregiver provides informed consent for themselves and their child to participate

Exclusion Criteria:

* none

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Child development | 10 months
  Child development measured using the Global Scales of Early Development - Long Form (GSED-LF). GSED-LF is based on direct administration by a research assistant. GSED-LF provides one score for the overall development of children 0-36 months of age. GSED scores will be age-standardized to a mean of 0 and a standard deviation of 1. Higher scores will indicate improved early developmental skills.

SECONDARY OUTCOMES:
Child socioemotional development | 10 months
  Child socioemotional development based on observational rating by a research assistant using an adapted version of the Wolke Scales (e.g., child affect, vocalization, cooperation with the research assistant). An average score will be calculated across the items with higher scores indicating more positive child behaviors.
Attitudes towards parenting | 10 months
  Primary caregivers will report the extent to which they agree with various statements about parental roles and engagement in nurturing care practices. A total score will be calculated with higher scores indicating more supportive parenting attitudes.
Caregiving environment | 10 months
  Caregiving environment will be assessed using the Home Observation for Measurement of the Environment for infants and toddlers aged 0 to 3 years (HOME-IT). It combines caregiver-reported items and observations of parenting behaviors to assess early learning opportunities at home and responsive caregiving behaviors of primary caregiver with the child. A total score will be calculated with higher scores indicate more responsive caregiving and enriched home learning environments.
Caregiver stimulation practices | 10 months
  Caregiver stimulation practices reported by primary caregiver about their engagement in early learning activities with the child (e.g. singing, telling stories). Activities adapted from the Family Care Indicators. A total score will be calculated with higher scores indicating more engagement in stimulation activities.
Caregiver disciplinary practices | 10 months
  Caregiver disciplinary practices reported by primary caregivers in terms of harsh punishment (e.g., shook the child, shouted at child) and positive disciplinary practices (e.g., explained why the behavior was wrong) used towards the child. Items adapted from Child Discipline Module of Multiple Indicator Cluster Survey. Separate indicators will be created for use of any harsh disciplinary practices or any positive disciplinary practices.
Infant and young child feeding practices | 10 months
  Infant and young child feeding (IYCF) practices including caregiver-reported breastfeeding and exclusive breastfeeding practices and child dietary diversity score (number of food groups the child consumed in previous 24 hours) based on WHO guidelines.
Parenting stress | 10 months
  Parenting distress reported by the primary caregiver using the Parenting Stress Index-Short Form, Parental Distress subscale. Higher total scores indicate greater parenting distress.
Depressive symptoms | 10 months
  Depressive symptoms reported by the primary caregiver using the Centre for Epidemiological Studies Depression Scale-10 items (CESD-10). Caregivers report on the frequency of depressive symptoms in the previous week. Items are summed to create an overall depression score, with higher scoring indicating greater depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Jeong, ScD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- B&M Consult, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalam MA, McCann JK, Shakil Z, Gambari A, Ochieng M, Jeong J. Maternal Mental Health and Child Dietary Diversity in Rural Kenya: Findings From a Pooled Analysis of 2 Baseline Studies. Curr Dev Nutr. 2025 Jun 24;9(7):107497. doi: 10.1016/j.cdnut.2025.107497. eCollection 2025 Jul. PMID 40718429
- [Derived] Jeong J, McCann JK, Onyango S, Ochieng M. A parenting program delivered through existing community-based peer groups to improve early child development in Homabay and Busia Counties, Kenya: study protocol for a cluster-randomized controlled trial. BMC Pediatr. 2024 Sep 17;24(1):592. doi: 10.1186/s12887-024-05065-7. PMID 39289646